CLINICAL TRIAL: NCT05765383
Title: Prognosis and Influencing Factors of Asthma in Children Aged 5-12 Years
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: ES-2023-005-01
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Asthma in Children
Keywords: prognosis; risk factors; phenotype; Persistent asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to 1)analyze the basic information of confirmed cases of asthma in children aged 5-12 years old hospitalized in the First Affiliated Hospital of Guangzhou Medical University from 2009 to 2020, 2)investigate the onset of asthma after 13 years old, 3)conducte lung function, blood and airway inflammation indicators, blood IL13 and IL1RL1 levels, 4)analyze the prognosis and influencing factors of children with asthma in this age group.Participants will be asked to fill a case report form and questionnaires. Besides, they should provide examination results like lung function, total IgE, expired nitric oxide, blood and sputum granulocyte counts, and determination of blood IL13 and IL1RL1 levels over the past 6 months.

DETAILED DESCRIPTION:
Research methods:

Part I: Retrospective analysis of hospitalized cases of asthma in children aged 5-12 years old from 2009 to 2020: (1) General information of the children (gender, age and BMI); (2) Special medical history of parents; (3) The history of respiratory virus infection in the early life; (4) that age of the first occurrence of asthma; (5) The number of wheezes in the 12 months before the diagnosis of asthma; (6) Specificity; (7) trigger factors of symptoms; (8) Time pattern of symptom manifestations; (9) Illness severity; (10) Airway inflammation pattern; (11) Baseline of lung function; (12) Anti-inflammatory treatment; (13) Reactions to drug therapy. (14) coinfected diseases or complications. (15) Genetic information.

Part II: Patients who are lost to follow-up will be excluded. The patients will be divided into asthma relief group and asthma continuation group according to whether they had relapsed asthma after 13 years old. The case report form and C-ACT/ACT questionnaire will be filled out. Patients should provide examination results like lung function, total IgE, expired nitric oxide, blood and sputum granulocyte counts, and determination of blood IL13 and IL1RL1 levels over the past 6 months.

Part III: Univariate and multivariate analyses will be performed for different prognostic outcomes of asthma in children aged 5 to 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized children with asthma (age range 5-12 years old) from 2009 to 2020 in the First Affiliated Hospital of Guangzhou Medical University were collected. Diagnostic criteria were included by referring to global initiative for asthma and Guidelines for Diagnosis, Prevention and Treatment of Pediatric Bronchial Asthma revised in 2008.

Exclusion Criteria:

* Children who declined follow-up
* Children with pulmonary and tracheal dysplasia, bronchiolitis obliterans, and other conditions leading to wheezing

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized children with asthma (age range 5-12 years old) from 2009 to 2020 in the First Affiliated Hospital of Guangzhou Medical University were collected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Review and collation. | 2022.08-2022.10
  To collect the case data of asthma in children aged 5 - 12 and analyze its clinical phenotype.
Case follow-up | 2022.10-2022.12
  The case report form and C-ACT/ACT questionnaire will be filled out. Patients should provide specific examination results.
Data analysis | 2023.1-2023.2
  Analyze the data obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China